CLINICAL TRIAL: NCT03625128
Title: Phase 0 Evaluation of Clinical and Neuroimage (18F-PM-PBB3 PET) Study in Tauopathy Including Alzheimer's Disease, Other Dementias and Normal Controls
Brief Title: 18F-PM-PBB3 PET Study in Tauopathy Including Alzheimer's Disease, Other Dementias and Normal Controls
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201700982A0
Record Dates: First submitted 2018-07-12; First posted 2018-08-10 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease; Cortical Basal Syndrome; Frontotemporal Dementia; Progressive Supranuclear Palsy; Vascular Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-18 PMPBB3 (Experimental): F-18 PMPBB3 imaging
  Interventions: Drug: F-18

INTERVENTIONS:
Drug: F-18 — This is an open-label study to evaluate the performance of a novel tau imaging ligand in up to 36 subjects (12 AD, 3 FTD, 3 PSP, 3 CBS, 3 VCI and 12 HV).
  Other Names: F-18 PMPBB3

SUMMARY:
This is an open-label study to evaluate the performance of a novel tau imaging ligand in up to 36 subjects (12 AD, 3 FTD, 3 PSP, 3 CBS, 3 VCI and 12 HV). Subjects will be recruited from the patient population and healthy volunteers of Taiwan residents. This study protocol requires each subject to complete the following components: screening evaluation, brain MRI and 18F-PM-PBB3 PET imaging up to two sessions. The screening procedures will include neuropsychological assessments, vital signs, ECG, physical examinations and laboratory tests. In addition, 18F-AV-45 PET imaging result will be as a part of inclusion criteria to confirm presence of amyloid deposition in patients with clinically diagnosed probable AD or absence of amyloid deposition in FTD, VCI and HV subjects. Furthermore, 18F-AV-133 PET imaging data will also be as a part of inclusion criteria to confirm the diagnosis of PSP and CBS. All subjects will complete clinical assessments and clinical safety tests to ensure the subject is medically stable to complete the study protocol. The screening procedures will occur within 30 days prior to 18F-PMPBB3 PET imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
3. Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
4. Male subjects must not donate sperm for the study duration.
5. Willing and able to cooperate with study procedures

Exclusion Criteria:

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes (except for patients with VCI), acute myocardial infarction, poorly controlled diabetes, previous head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases.
3. Current or prior history of major psychiatric disorders, epilepsy and major depression.
4. History of severe allergic or anaphylactic reactions particularly to the tested drugs.
5. History of positive test for human immunodeficiency virus (HIV).
6. Life expectancy less than 1 year.
7. Pregnant women, lactating or breast-feeding women.
8. Clinically significant abnormal laboratory values and/or clinically significant or unstable medical or psychiatric illness.
9. Substance abuse or alcoholism for at least 3 months.
10. Cognitive impairment resulting from trauma brain injury.
11. Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv.
12. Subject has received an investigational drug or device within 30 days of screening
13. Patients in whom MRI was contraindicated and with history of claustrophobia in MRI
14. General MRI, and / or PET exclusion criteria. MRI exclusion criteria include: Findings of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension, except for patients with VCI), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
15. Severe language impairment precluding cognitive assessments, defined as a score of 3 points in the language score of the National Institute of Health Stroke Scale.
16. Subjects having high risks for the study according to the PI discretion.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are to evaluate the dosimetry of novel radiotracer 18F-PM-PBB3 in human. | YEAR ONE
  Time-integrated activity in each organ will be calculated by trapezoidal integration of the first 45 min of the organ's time-activity curve, followed by a single-exponential fit to the remaining data points (based on the 4 whole-body images) extrapolate to infinity, all base on non-decay-corrected data.Residence times will be obtained by dividing the time-integrated activity by the injected amount of activity.

SECONDARY OUTCOMES:
Optimal scanning time for brain imaging using 18F-PM-PBB3 . | YEAR ONE
  PET data will be acquired using SIMENS PET/CT or PET/MRI scanner with an axial field of view of 15.7cm. For PET/CT protocol, a 50-min dynamic brain PET scan (6x10s, 4x60s, 5x180s, 6x300s) will be started simultaneously with the injection of 10mCi of 18F-PM-PBB3 after a low-dose CT scan for patient positioning and attenuation correction.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chang Huang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan, Guishan Dist, Taiwan

REFERENCES:
- [Derived] Lin KJ, Huang SY, Huang KL, Huang CC, Hsiao IT. Human biodistribution and radiation dosimetry for the tau tracer [18F]Florzolotau in healthy subjects. EJNMMI Radiopharm Chem. 2024 Apr 2;9(1):27. doi: 10.1186/s41181-024-00259-x. PMID 38563872